CLINICAL TRIAL: NCT01883245
Title: Effects of Transcranial Direct Current Stimulation (tDCS) in Patients With Chronic Orofacial Pain Unresponsive to Conventional Treatment. A Randomized Controlled Trial.
Brief Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Patients With Chronic Orofacial Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: We decided to stopped the study because we have difficulties in recruiting subjects phase.
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, MD, MD, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Orofacial pain_tDCS
Record Dates: First submitted 2013-06-18; First posted 2013-06-21 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-01

CONDITIONS: Orofacial Pain
Keywords: Orofacial chronic pain; tDCS; Transcranial direct current stimulation; Brain stimulation
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sham tDCS (Active Comparator): This group will receive sham-tDCS for 5 days. The anode will be placed on the primary motor cortex (M1) of the dominant hemisphere and the cathode on the contralateral supraorbital area. The direct current is transmitted through a pair of sponge electrodes, with a surface of 35 cm2 (7x5), soaked in saline solution and, it is generated by a constant current stimulator, with rechargeable batteries. This continuous stimulation lasted 30 seconds, with an intensity of 1 milliampere.
  Interventions: Device: sham tDCS
- real tDCS (Experimental): This group will receive continuous stimulation lasting 20 minutes daily, for 5 days.
  Transcranial direct current stimulation (tDCS) will be administered as follows. The anode will be placed on the primary motor cortex (M1) of the dominant hemisphere and the cathode on the contralateral supraorbital area. The direct current is transmitted through a pair of sponge electrodes, with a surface of 35 cm2 (7x5), soaked in saline solution and, it is generated by a constant current stimulator, with rechargeable batteries. This continuous stimulation lasted 20 minutes, with an intensity of 1 milliampere.
  Interventions: Device: real tDCS

INTERVENTIONS:
Device: real tDCS — 2 milliampere real direct current stimulation for 20 minutes daily for 5 days.
  Arms: real tDCS
Device: sham tDCS — 2 milliampere sham direct current stimulation for 20 minutes daily for 5 days.
  Arms: sham tDCS

SUMMARY:
Patients affected by chronic orofacial pain represent an emergent medical problem due to the lack of knowledge on the cause, pathophysiology and psychology of many of these conditions, that belongs to a multifactorial origin.

Particularly, temporomandibular joint disorders involve a series of symptoms that refers both to intrinsic and extrinsic joint conditions where pain can be associated to a reduction of the joint movement, click or to other sounds of the joint.

The lack of a recognized causal therapy led to the suggestion of many treatment modalities with a multidisciplinary approach for the management of symptoms that include the use of occlusal splints, physiotherapy-speech therapy, behavioral and physical therapy, drugs, chirurgical approaches. In most cases these strategies together allow the control of the symptoms, even though they aren't completely resolutive.

In these patients is frequent chronic pain and ineffectiveness of common drugs used.

It has been demonstrated how transcranial electrical brain stimulation with direct current (tDCS) is able to reduce the intensity and the duration of chronic pain.

Stimulating the motor cortex can reduce pain by modulating brain activities in the areas involved in cerebral circuits controlling pain, such as thalamus, facilitating the descendant inhibitory mechanisms and enhancing the number of opiates receptors.

This clinical trial is based on the evaluation of the effects of tDCS on pain and on activities daily living (ADL) participation patients with chronic orofacial pain that don't respond to other treatments.

DETAILED DESCRIPTION:
Inclusion criteria:

* Male and female between 18 and 75 years old
* Clinic history of previous orofacial and/or dental surgery
* Chronic orofacial pain for more than a year measurable by the VAS more than 3 .
* Pain not responsive to pharmacological treatment (analgesic, anti inflammatory, opiaces, antidepressant drugs and physiotherapy modalities)

Outcome measures:

Subjects will be assessed before the beginning of the treatment (T0), after tDCS (T1) and after one month of stimulation(T2) .

In the two weeks prior to T0 the patient will be asked in a questionnaire to report daily the level of pain, anxiety and state of mind using the VAS. This period of observation is necessary for the patient to get used to these measures and to underline possible intra-subject changing.

• Clinic scales

-Visual Analogue Scale (VAS): it is one of the most used between scales for pain evaluation [18]

RDC/TMD AXIS I: diagnostic classification for temporomandibolar disfunction. RDC/TMD AXIS II: behavioral questionnaire (7 questions about chronic pain severity) which evaluates chronic pain following the graded scale for chronic pain.

* Symptoms Checklist-90-R scales (SCL 90-R): Depression and anxiety assessment for non-specific physical symptoms
* electrical pain threshold: The Digitimer High Voltage Stimulator model DS74 provides high voltage pulses of constant current up to 100mA, pulses are of short duration and the output current is variable ranging between 0 and 100mA. The Digitimer is used to evaluate the pain perception threshold by applying electrical stimulation to the index finger to a pulse duration of 200 ls. The initial current applied is 0mA and increases of 0.1 mA until the subject feels pain.
* Oral Health Impact Profile 49 (OHIP 49): provides a measure of social impact of oral disorders by providing a comprehensive measure of dysfunction, discomfort and disability resulting from the oral cavity conditions. The OHIP-49 is based on the adaptation of the World Health Organization classification.
* Pain detect Questionnaire

Pressor pain threshold

ELIGIBILITY:
Inclusion Criteria:

* Male and female between 18 and 75 years old
* Clinic history of previous orofacial and/or dental surgery
* Chronic orofacial pain for more than a year measurable by the VAS more than 3 .
* Pain not responsive to pharmacological treatment (analgesic, anti inflammatory, opiates, antidepressant drugs and physiotherapy modalities)

Exclusion Criteria:

* Contraindication to tDCS: presence of metallic implants that can be stimulated, moved or overheated by electric current, positive anamnesis for epilepsy, implantable systems ( ventriculoperitoneal shunt, pacemaker, intracranial pumps, intracranial metallic systems)
* Major neurological or psychiatric pathologies
* Pregnancy
* Severe hepatorenal and cardiopulmonary diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Visual Analogue Scale (VAS) for pain | 1) one day pre-tDCS 5 days treatment. 2) Every day, for 5 days pre and post tDCS stimulation. 3) one day post tDCS 5 days treatment. 4)Follow up at one month.
  Visual analogue scale measure for pain. Score range from 0-10. For rating overall pain: mild = 1-3, moderate = 4-7, severe = 8-10 For rating Chronic Pain, excellent internal consistency for a single pair of rating between Numeric Pain Rating Scale and Visual Analogue Scale (r = 0.86)

SECONDARY OUTCOMES:
Research Diagnostic Criteria Temporomandibular disorders (RDC/TMD) AXIS I | 1) one day pre 5 days tDCS treatment. 2) one day post 5 days tDCS treatment 3) One month follow up
  Diagnostic classification for temporomandibular disfunction.
Research Diagnostic Criteria Temporomandibular disorders RDC/TMD AXIS II | 1) one day pre 5 days tDCS treatment. 2) one day post 5 days tDCS treatment 3) One month follow up
  Behavioral questionnaire (7 questions about chronic pain severity) which evaluates chronic pain following the graded scale for chronic pain.
Symptoms Checklist 90-R scales (SCL 90-R) | 1) one day pre 5 days tDCS treatment. 2) one day post 5 days tDCS treatment 3) One month follow up
  Depression and anxiety assessment for non-specific physical symptoms.
Electrical and pressure pain threshold | 1) one day pre 5 days tDCS treatment. 2) one day post 5 days tDCS treatment 3) One month follow up
  The device for assessing pain is a high voltage stimulator provides high voltage pulses of constant current up to 100 milliampere, pulses are of short duration and the output current is variable ranging between 0 and 100 milliampere. This device is used to evaluate the pain perception threshold by applying electrical stimulation to the index finger to a pulse duration of 200 ls. The initial current applied is 0 milliampere and increases of 0.1 milliampere until the subject feels pain.
Oral Health Impact Profile 49 (OHIP 49) | 1) one day pre 5 days tDCS treatment. 2) one day post 5 days tDCS treatment 3) One month follow up
  Provides a measure of social impact of oral disorders by providing a comprehensive measure of dysfunction, discomfort and disability resulting from the oral cavity conditions. The OHIP-49 is based on the adaptation of the World Health Organization classification.
Pain detect Questionnaire (PD-Q) | 1) one day pre 5 days tDCS treatment. 2) one day post 5 days tDCS treatment 3) One month follow up
  The PD-Q is a reliable screening tool with high sensitivity, specificity and positive predictive accuracy.
  Simple, patient-based, easy-to-use screening questionnaires can determine the prevalence of neuropathic pain components both in individual low back pain patients and in heterogeneous cohorts of such patients. Since NeP correlates with more intense pain, more severe co-morbidity and poorer quality of life, accurate diagnosis is a milestone in choosing appropriate therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ferrara University Hospital, Ferrara, Ferrara, Italy